CLINICAL TRIAL: NCT04855084
Title: Occlusal Relationship Assesment of Monolithic Zirconia Fixed Dental Prosthesis
Brief Title: Occlusal Relationship Assesment of Monolithic Zirconia FDPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duygu Karasan (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Duygu Karasan, Research Asistant, DDS, PhD, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA-180043
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Tooth-loss
Keywords: Occlusal Relationship; Complete Digital Work-flow; Fixed Partial Denture; Fixed Dental Prosthesis
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Intervention Model Description: A non-randomized one-control group study
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Complete Digital Fixed Dental Prosthesis (Experimental): Following the Digital Impression using 3 Shape Trios Intraoral scanner, digital design, and manufacturing of the Monolithic Zirconia FDPs.
  Monolithic FDPs: before adjustment
  Using Intraoral Scanner, occlusal relationship assessment of the Monolithic FDPs before the occlusal adjustment.
  Monolithic FDPs: after adjustment
  Using Intraoral Scanner, occlusal relationship assessment of the Monolithic FDPs after the occlusal adjustment.
  Interventions: Other: Monolithic FDPs: before adjustment; Other: Monolithic FDPs: after adjustment; Other: Metal fused porcelain FDPs: before adjustment; Other: Metal fused porcelain FDPs: after adjustment
- Analog Fixed Dental Prosthesis (Active Comparator): Following the Conventional Impression, transfer to the articulator with Face bow. Manufacturing of the FDPs with lost wax technique and veneering.
  Metal fused porcelain FDPs: before adjustment
  Using Intraoral Scanner, occlusal relationship assessment of the metal fused to porcelain FDPs before the occlusal adjustment.
  Metal fused porcelain FDPs: after adjustment
  Using Intraoral Scanner, occlusal relationship assessment of the metal fused to porcelain FDPs after the occlusal adjustment.
  Interventions: Other: Monolithic FDPs: before adjustment; Other: Monolithic FDPs: after adjustment; Other: Metal fused porcelain FDPs: before adjustment; Other: Metal fused porcelain FDPs: after adjustment

INTERVENTIONS:
Other: Monolithic FDPs: before adjustment — Before the occlusal adjustment, Occlusal relationship recording of the 3-unit monolithic FDPs which was fabricated following the complete digital work-flow.
Other: Monolithic FDPs: after adjustment — After the occlusal adjustment, Occlusal relationship recording of the 3-unit monolithic FDPs which was fabricated following the complete digital work-flow.
Other: Metal fused porcelain FDPs: before adjustment — Before the occlusal adjustment, Occlusal relationship recording of the 3-unit metal fused porcelain FDPs which was fabricated following the complete conventional manufacturing procedure.
Other: Metal fused porcelain FDPs: after adjustment — After the occlusal adjustment, digital occlusal relationship recording was done of the 3-unit metal fused porcelain FDPs which was fabricated following the complete conventional manufacturing procedure.

SUMMARY:
To analyze in vivo occlusal accuracy and occlusal adjustment requirement, a cross-over clinical trial was designed. Two 3-unit tooth-supported posterior FDPs were planned to be made for each patient's single missing tooth gap, one with complete analog workflow (control group) and the other complete digital workflow (test group). The analog workflow aims for a porcelain fused to metal (PFM) FDP whereas the digital workflow aims for 3-unit monolithic Zr FDP. PFor half of the restorations, digital impression was planned to be taken first and to be followed by analog impression. As for the occlusal adjustment, in half of the study sites monolithic Zr FDPs were planned to be tried-in first, followed by metal-ceramic FDP and vice versa.

One investigator (DK) was assigned to prepare the restoration sites and deliver the FDPs. All monolithic Zr and all metal-ceramic FDPs were designed and fabricated by the same experienced dental technician. One investigator (HL), that was not involved in the treatment intervention was assigned to make the 3D analysis of the volumetric occlusal adjustment amount.

DETAILED DESCRIPTION:
All teeth preparations will be carried out ensuring the minimum material thickness for monolithic FDPs (0.8-1 mm margin thickness, 1 mm occlusal thickness) by one experienced investigator (DK). To prevent any possible carry-over effect, the impression acquisition order will be randomized.

The control group FDPs (metal-ceramic) will be fabricated with a complete analog workflow. Accordingly, a polyether dual-phase impression (Impregum Penta Soft Quick and Soft Quick, 3M) will be taken from the restoration arch and a Polyvinylsiloxane (PVS) impression material will be used for the impression of the antagonist arch. Face bow transfer (Whip Mix Face bow0 will be done. Following the stone master model (Type IV dental rock, Fuji) obtention, the maxillary models will be mounted to a semi-adjustable articulator based on the face bow record and mandibular models will be then mounted with the aid of laterotrusive and MI records. The MI and laterotrusive records will be taken with a PVS bite registration material. The Cr-Ni frameworks will be fabricated with lost-wax technique (Brand?), manually layered with feldspathic veneering porcelain (Vita), and glazed by one experienced dental technician.

The test group FDPs (high translucent monolithic Zr) (Aidite Multilayer 3D) will be fabricated by a complete/model-free digital workflow. The digital quadrant impressions of the preparation, antagonist as well as bite registration will be obtained by the use of an IOS (Trios 3, 3Shape). The files will be sent to a CAD software (Dental System, 3Shape) directly via the communication tool (3 Shape Communicate, 3Shape). Following CAD, the high translucent monolithic Zr 3-unit FDPs will be computer-aided manufactured (CORITEC 350i Loader, imes-icore GmbH). FDPs will be high-gloss polished, glazed, and sent to the dental clinic for the try-in session. Monolithic Zr design and manufacturing process will be completed by one dental technician that is highly experienced in CAD/CAM.

Clinical occlusal adjustment:

A standardized occlusal adjustment strategy will be adopted and executed by one investigator for both control and test group FDPs. In half of the restoration sites, monolithic Zr restorations will be the ones to have been tried first whereas in the other half metal-ceramic FDPs were the first. Initially, distal and mesial approximal contact areas, then the internal fit will be checked and adjusted to eliminate any interferences in order to ensure the optimal fitting of the restorations. For the occlusal adjustment amount calculation, the FDPs will be fixed on the prepared teeth provisionally and scanned by an IOS (Trios 3, 3Shape) to record the pre-adjustment FDP volume. The occlusal contacts and adjustment needs were assessed while still the restorations are fixed. The occlusal adjustment strategy will be as follows: Under normal occlusal forces, 40-micron articulation paper (Arti-Check micro-thin, Bausch, Cologne, Germany) will be used and followed by 12-micron articulation foil (Shimstock-foil, Bausch, Cologne, Germany) under strong occlusal force. The FDPs' occlusal contact design will be ensured to hold the articulation foil under strong occlusal force. Thereafter, once ensuring the FDPs to remain fixed, intraoral digital quadrant impressions (Trios 3, 3 Shape) will be taken by the same investigator in order to record the post-adjustment volume of the FDPs. After chairside finishing and polishing of the adjustment areas, Monolithiz Zr FDPs will be adhesively luted by a composite cement as the definitive restoration.

2.4. Quantitative analysis Both .stl files (pre-and-post adjustment) will be exported in order to process in an inspection software (Gom Inspect 2019, GOM GmbH, Braunschweig, Germany). The pre-and post-adjustment .stl files will be superimposed with the surface of restorations excluding occlusal adjusted area. After that, they will be sectioned from the same planes, mesial, distal, and 3mm apical to occlusal plane. The total volume of the sections that will be analyzed will be measured and the quantitative volume difference of the sectioned parts then was Calculated three-dimensionally (3Matic, Materialise NV, Leuven, Belgium). The total volumetric difference in mm3 between pre-and post-adjustment .stl files will be calculated for each 3-unit FDP

ELIGIBILITY:
Inclusion Criteria for the participants:

1. The individuals with the mandibular or maxillary single missing occlusal unit (2nd premolar, 1st molar) adjacent to a premolar and/or molar tooth
2. Participants over 20 years old with no contradiction of dental treatment.
3. Good oral hygiene habits, healthy periodontal status, no sign of bruxism (e.g. attrition score >2 according to Wigdorowicz-Makowerowa, and/or muscle pain), and no self-reported grinding and/or clenching.

Inclusion criteria for the abutment teeth included:

1. No visible periapical lesion
2. Presence of minimum 1:1 crown/root ratio
3. Class I mobility (Nyman & Lindhe 2003)
4. No probing depth more than 4mm
5. Presence of natural opposing teeth with no restorative treatment.
6. Presence of a stable maximum intercuspation (MI) relationship

Exclusion Criteria:

* Patients and teeth that are not fulfilling the inclusion criteria

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
The evaluation of effectiveness of workflows by assesing the occlusal registration accuracy of 3-unit FDPs that were fabricated with two different work-flows | At the baseline, the same day of delivery
  The occlusal registration accuracy and effectiveness of both analog and digital workflows by means of comparing quantitatively the occlusal adjustment requirement of 3-unit tooth supported metal-ceramic and Zr FDPs produced by analog work-flow use of semi-adjustable articulators with face-bow transfer and complete digital workflow, respectively

SECONDARY OUTCOMES:
Operator and Patient reported outcomes | Impression visit and baseline visit (restoration delivery)
  The patient and operator reported outcomes will be evaulated by means of visual analog scales (VAS). The patients and operator will be asked to rate from 0 to 10 their experience of impression and overall treatment procedure.
  (0: inconvenient, 10 very convenient)

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Karasan, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Dentistry, Ankara, Turkey (Türkiye)